CLINICAL TRIAL: NCT02382484
Title: Impact of Pacing Site and AV Delay on Blood Pressure in Hypertensive Patients: An Acute Study in Patients Undergoing an Electrophysiology Study or Pacemaker Implant
Brief Title: Impact of Pacing Site and AV Delay on Blood Pressure in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BackBeat Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acute FIM Study - China
Record Dates: First submitted 2015-02-18; First posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension
Keywords: Hypertension Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension; Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): The study was a single arm, unblinded, treatment only study. Each patient served as his or her own control.
  Treatment delivered by a dual chamber pacing system (BackBeat Medical) which was able to generate stimulating patterns with characteristics that are different than the common pacemaker.
  The study was limited to hypertensive patients who were also already scheduled to undergo an invasive electrophysiology procedure.
  Interventions: Device: A dual chamber pacing system (BackBeat Medical)

INTERVENTIONS:
Device: A dual chamber pacing system (BackBeat Medical) — For each patient, one pacing electrode was placed in the right atrium and the second electrode was placed in the right ventricle. With a dual chamber pacing system (BackBeat Medical) it was possible to pace the heart with a wide variety of pacing settings.

SUMMARY:
The purpose of this study is to test whether the A-V sequential pacing strategy shown to effectively reduce blood pressure in a dog model of hypertension also reduces blood pressure acutely in patients with hypertension (systolic blood pressure greater than 140 mmHg) despite medical treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has hypertension with systolic blood pressure >140 mmHg despite at least one antihypertensive medication.
2. Patient has a clinical indication for a pacemaker or an electrophysiology study involving introduction of transvenous electrophysiology catheters to the right atrium and/or right ventricle.
3. Patient is willing and able to provide informed consent

Exclusion Criteria:

1. Patient is in atrial fibrillation at the time of the study
2. Patient has an ejection fraction less than 45%
3. Patient has a history of symptomatic heart failure, regardless of EF
4. Patient is undergoing an ablation procedure for a bypass track (WPW)
5. Patient has a history of resuscitation from ventricular fibrillation or sustained ventricular tachycardia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change of blood pressure upon initiation of pacing with AV delays of 2 ms | Approx. 5 minutes after initiating pacing with the respective AV delay
Change of blood pressure upon initiation of pacing with AV delays of 20 ms | Approx. 5 minutes after initiating pacing with the respective AV delay
Change of blood pressure upon initiation of pacing with AV delays of 40 ms | Approx. 5 minutes after initiating pacing with the respective AV delay
Change of blood pressure upon initiation of pacing with AV delays of 80 ms | Approx. 5 minutes after initiating pacing with the respective AV delay
Assessment of any adverse effects | Over a 24 hour period following the acute tests

CONTACTS AND LOCATIONS:
Overall Officials: Bing Yang, MD, Principal Investigator — The Department of Cardiology, The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- The Department of Cardiology, The First Affiliated Hospital of Nanjing Medical University, Nanjing, China